CLINICAL TRIAL: NCT03163095
Title: Closed Versus Open Abdomen in the Surgical Treatment of Severe Secondary Peritonitis: a Randomized Controlled Clinical Trial
Brief Title: Closed or Open Abdomen for the Management of Abdominal Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Andrew W Kirkpatrick, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB16-1588-the COOL study
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Abdominal Sepsis; Abdominal Infection
Keywords: sepsis; abdominal infection; open abdomen management; Negative pressure peritoneal therapy
MeSH Terms: conditions — Intraabdominal Infections; Sepsis

STUDY DESIGN:
Intervention Model Description: Randomization by blocks on a website.
Who Masked: Outcomes Assessor
Masking Description: Research members in the laboratory will be blinded with participants' clinical data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Abdomen Management with ANPPT dressing (Active Comparator): The abdominal fascia will not be closed, but a temporally abdomenal closure (TAC) dressing (such as AbThera dressing) will be placed to protect the viscera with active Negative Pressure Peritoneal drain. Formal abdominal closure or dressing change at 24-72 hours from placement should be performed.
  Interventions: Device: Open Abdomen Management with ANPPT dressing
- Closed Abdomen Management (Sham Comparator): Primary closure of the abdominal fascia with placement of an intra-peritoneal drain (such as a Jackson-Pratt drain). Any decision to perform a re-laparotomy will be at the discretion of the treating surgical team.
  Interventions: Other: Closed Abdomen Management

INTERVENTIONS:
Device: Open Abdomen Management with ANPPT dressing — The abdominal fascia will not be closed, but a temporally abdominal closure (TAC) dressing, such as AbThera dressing, will be placed to protect the viscera with active Negative Pressure Peritoneal Therapy.
  The time that the TAC dressing will be changed will be left to the discretion of the attending surgeon, but practice guidelines mandate either formal abdominal closure or dressing change at 24-72 hours from placement.
  Blood samples and peritoneal fluid will be drawn up to 72 hours after enrollment.
  Arms: Open Abdomen Management with ANPPT dressing
Other: Closed Abdomen Management — Primary closure of the abdominal fascia with placement of an intra-peritoneal drain (such as a Jackson-Pratt drain).
  This strategy will allow drainage of intra-peritoneal fluid for both clinical reasons and to facilitate intra-peritoneal fluid testing. Closure or not of the skin will be left to the attending surgeons discretion. Any decision to perform a relaparotomy (Relaparotomy on Demand) will be at the discretion of the treating critical care teams, and in no way mandated by this recruitment.
  Blood samples and peritoneal fluid (if available) will be drawn up to 72 hours after enrollment.
  Arms: Closed Abdomen Management

SUMMARY:
This is a prospective randomized clinical study. The study will comprise the randomized decision to either A) primarily close the fascia after laparotomy for intra-abdominal infection (CLOSED); or B) leave the fascia open after laparotomy and apply a temporary abdominal closure (TAC) device (OPEN) with a vacuum drain.

Although debatable, both procedures (CLOSED or OPEN abdomen) are acceptable based on current suggested standard of care. Thus, high quality data to direct clinical decision making in this highly lethal condition is urgently required.

DETAILED DESCRIPTION:
Severe complicated intra-abdominal sepsis (SCIAS) is a World-Wide challenge, with high mortality rates, and ever increasing incidence. Most cases are subjected to secondary peritonitis in which there is a physical disruption of the integrity of the gastrointestinal (GI) tract leading to contamination of the peritoneal cavity. Ultimately, the resultant organ damage results in auto-amplifying biomediator generation and systemic inflammation. Mortality rates range from 10% to over 40% when shock is present. The key principles of treating SIAS are early antibiotic administration and the earliest possible operative intervention to provide source control of GI perforations/disruptions. A further potential therapeutic option may be to utilize open abdomen (OA) management with active negative peritoneal pressure therapy (ANPPT) to remove intra-peritoneal inflammatory ascites and to ameliorate the systemic damage from SCIAS. Recent data from a randomized controlled trial including either severe peritonitis or trauma patients, showed the 30-days mortality differed between commercial open abdomen systems and non-commercial technique, which favored the more effective commercial device. Although there is a biologic rationale for such an intervention from animal models as well as non-standardized clinical utilization currently, the open abdomen management with ANPPT remains a novel therapy with much clinical equipoise. Thus, the Closed Or Open after Laparotomy (COOL) study will constitute a prospective randomized controlled trial to address this issue.

There is a complex relationship between pressure, ischemia, and inflammation within the peritoneal cavity. Independently the damaged gut seems to act as a continued source of inflammation propagating systemic inflammatory response syndrome (SIRS) and potentiating multi-organ dysfunction syndrome (MODS). Although extremely complicated, visceral ischemia further generates multiple immunological mediators with the pro-inflammatory cytokines tumor necrosis factor-alpha (TNF-α), and interleukin 6 (IL-6), as well as inhibitive cytokines such as interleukin 10 (IL-10). Post-operative complications associate with increasing levels of systemic IL-6, and peritoneal TNF-α. Jansson and colleagues believe that peritoneal cytokines in humans respond more extensively compared to systemic cytokines, and that a normal postoperative course is characterized by decreasing levels of peritoneal cytokines based on studies of both elective and emergency surgery. Overall, the peritoneal cytokine response is much higher than the systemic response in peritonitis.

ANPPT therapy may be a more direct and focused solution to this complicated problem, and that will be complementary to the other benefits of open abdomen management in the sickest patients. Whether improved post-operative courses can be obtained through this relatively simple approach of actively removing peritoneal cytokines in humans is therefore a secondary objective of this trial.

Another potential benefit of ANPPT after severe infection may be the attendant decompression of the abdominal compartment and prevention of even modest degrees of intra-abdominal hypertension (IAH). Patients with intra-abdominal infections are at risk of elevated intra-abdominal pressure (IAP) both as a result of the primary intra-peritoneal disease, and as large fluid resuscitation often required maintaining organ perfusion. Recent studies have demonstrated a high prevalence of IAH following aggressive resuscitation of septic patients. Intra-abdominal hypertension is present in as many as 80% of septic medical and surgical ICU patients. Reintam also reported that septic patients with IAH had a 50% rate of mortality compared to 19% without IAH, making IAH a significant marker for an increased risk of death. Within our own institution, rates of IAH were over 87% of septic ICU patients and further 61% of these patients had severe IAH at levels commensurate with abdominal compartment syndrome (ACS). Although direct translation to humans is uncertain, even modest degrees of IAH (often clinically ignored) have been found to have profound effects on propagating multiple organ failure in animals with ischemia/intra-peritoneal infections.

The study intervention will comprise the randomized decision to either A) primarily close the fascia after laparotomy for SCIAS (CLOSED); or B) leave the fascia open after laparotomy for SCIAS and apply an ANPPT temporary abdominal closure (TAC) device (OPEN).

Patients will be randomized intra-operatively once it is determined that COMPLICATED and SEVERE Intra-Abdominal Infection (SCIAS) is present. SEVERE will be defined and denoted by the presence of any organ dysfunction exemplified by septic shock OR a Predisposition-Infection-Response-Organ Dysfunction Score > 3 or a World-Society-of-Emergency-Surgery-Sepsis-Severity-Score > 8, and COMPLICATED with the presence of purulent, feculent, or enteric spillage over at least 2 intra-peritoneal quadrants.

ELIGIBILITY:
Inclusion Criteria:

* Presence of purulent, feculent, or enteric spillage over at least 2 intra-peritoneal quadrants intra-operatively;
* Septic shock, or
* Predisposition-Infection-Response-Organ Dysfunction Score > 3, or
* World-Society-of-Emergency-Surgery-Sepsis-Severity-Score > 8

Exclusion Criteria:

* Pregnant;
* Confirmed or strongly suspected severe IAH (IAP>20 mmHg);
* No intentional of providing ongoing care;
* pancreatitis as the source of peritonitis;
* uncontrolled bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2019-06-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The numbers of participants who are survival in hospital stay | 90 days after participants enrolled in the study
  The rate of survival of participants in both arms

SECONDARY OUTCOMES:
The days of intensive care unit stay | 30 days after participants enrolled in the study
  The median length of days in ICU needed by participants in both arms
The pg/ml of blood Interleukin-6 | 72 hours after participants enrolled in the study
  The mean concentrations of blood IL-6 in participants in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Kirkpatrick, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Not shared.

REFERENCES:
- [Background] Kirkpatrick AW, Sugrue M, McKee JL, Pereira BM, Roberts DJ, De Waele JJ, Leppaniemi A, Ejike JC, Reintam Blaser A, D'Amours S, De Keulenaer B, Malbrain MLNG. Update from the Abdominal Compartment Society (WSACS) on intra-abdominal hypertension and abdominal compartment syndrome: past, present, and future beyond Banff 2017. Anaesthesiol Intensive Ther. 2017;49(2):83-87. doi: 10.5603/AIT.a2017.0019. Epub 2017 May 14. No abstract available. PMID 28502071
- [Result] Xiao Z, Wilson C, Robertson HL, Roberts DJ, Ball CG, Jenne CN, Kirkpatrick AW. Inflammatory mediators in intra-abdominal sepsis or injury - a scoping review. Crit Care. 2015 Oct 27;19:373. doi: 10.1186/s13054-015-1093-4. PMID 26502877
- [Result] Kirkpatrick AW, Roberts DJ, Faris PD, Ball CG, Kubes P, Tiruta C, Xiao Z, Holodinsky JK, McBeth PB, Doig CJ, Jenne CN. Active Negative Pressure Peritoneal Therapy After Abbreviated Laparotomy: The Intraperitoneal Vacuum Randomized Controlled Trial. Ann Surg. 2015 Jul;262(1):38-46. doi: 10.1097/SLA.0000000000001095. PMID 25536308
- [Result] Kubiak BD, Albert SP, Gatto LA, Snyder KP, Maier KG, Vieau CJ, Roy S, Nieman GF. Peritoneal negative pressure therapy prevents multiple organ injury in a chronic porcine sepsis and ischemia/reperfusion model. Shock. 2010 Nov;34(5):525-34. doi: 10.1097/SHK.0b013e3181e14cd2. PMID 20823698
- [Result] Opal SM, Dellinger RP, Vincent JL, Masur H, Angus DC. The next generation of sepsis clinical trial designs: what is next after the demise of recombinant human activated protein C?*. Crit Care Med. 2014 Jul;42(7):1714-21. doi: 10.1097/CCM.0000000000000325. PMID 24717456
- [Result] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399
- [Result] Reintam A, Parm P, Kitus R, Kern H, Starkopf J. Primary and secondary intra-abdominal hypertension--different impact on ICU outcome. Intensive Care Med. 2008 Sep;34(9):1624-31. doi: 10.1007/s00134-008-1134-4. Epub 2008 May 1. PMID 18446319
- [Result] Regueira T, Bruhn A, Hasbun P, Aguirre M, Romero C, Llanos O, Castro R, Bugedo G, Hernandez G. Intra-abdominal hypertension: incidence and association with organ dysfunction during early septic shock. J Crit Care. 2008 Dec;23(4):461-7. doi: 10.1016/j.jcrc.2007.12.013. Epub 2008 Apr 18. PMID 19056007
- [Result] Malbrain ML, Chiumello D, Pelosi P, Wilmer A, Brienza N, Malcangi V, Bihari D, Innes R, Cohen J, Singer P, Japiassu A, Kurtop E, De Keulenaer BL, Daelemans R, Del Turco M, Cosimini P, Ranieri M, Jacquet L, Laterre PF, Gattinoni L. Prevalence of intra-abdominal hypertension in critically ill patients: a multicentre epidemiological study. Intensive Care Med. 2004 May;30(5):822-9. doi: 10.1007/s00134-004-2169-9. Epub 2004 Feb 3. PMID 14758472
- [Result] De Waele JJ. Abdominal Sepsis. Curr Infect Dis Rep. 2016 Aug;18(8):23. doi: 10.1007/s11908-016-0531-z. PMID 27363829
- [Result] Leppaniemi A, Kimball EJ, De Laet I, Malbrain ML, Balogh ZJ, De Waele JJ. Management of abdominal sepsis--a paradigm shift? Anaesthesiol Intensive Ther. 2015;47(4):400-8. doi: 10.5603/AIT.a2015.0026. Epub 2015 May 14. PMID 25973662
- [Result] Tellor B, Skrupky LP, Symons W, High E, Micek ST, Mazuski JE. Inadequate Source Control and Inappropriate Antibiotics are Key Determinants of Mortality in Patients with Intra-Abdominal Sepsis and Associated Bacteremia. Surg Infect (Larchmt). 2015 Dec;16(6):785-93. doi: 10.1089/sur.2014.166. Epub 2015 Aug 10. PMID 26258265
- [Result] Tolonen M, Sallinen V, Mentula P, Leppaniemi A. Preoperative prognostic factors for severe diffuse secondary peritonitis: a retrospective study. Langenbecks Arch Surg. 2016 Aug;401(5):611-7. doi: 10.1007/s00423-016-1454-8. Epub 2016 May 30. PMID 27241334
- [Result] Sartelli M, Viale P, Catena F, Ansaloni L, Moore E, Malangoni M, Moore FA, Velmahos G, Coimbra R, Ivatury R, Peitzman A, Koike K, Leppaniemi A, Biffl W, Burlew CC, Balogh ZJ, Boffard K, Bendinelli C, Gupta S, Kluger Y, Agresta F, Di Saverio S, Wani I, Escalona A, Ordonez C, Fraga GP, Junior GA, Bala M, Cui Y, Marwah S, Sakakushev B, Kong V, Naidoo N, Ahmed A, Abbas A, Guercioni G, Vettoretto N, Diaz-Nieto R, Gerych I, Trana C, Faro MP, Yuan KC, Kok KY, Mefire AC, Lee JG, Hong SK, Ghnnam W, Siribumrungwong B, Sato N, Murata K, Irahara T, Coccolini F, Segovia Lohse HA, Verni A, Shoko T. 2013 WSES guidelines for management of intra-abdominal infections. World J Emerg Surg. 2013 Jan 8;8(1):3. doi: 10.1186/1749-7922-8-3. PMID 23294512
- [Result] Sartelli M, Abu-Zidan FM, Catena F, Griffiths EA, Di Saverio S, Coimbra R, Ordonez CA, Leppaniemi A, Fraga GP, Coccolini F, Agresta F, Abbas A, Abdel Kader S, Agboola J, Amhed A, Ajibade A, Akkucuk S, Alharthi B, Anyfantakis D, Augustin G, Baiocchi G, Bala M, Baraket O, Bayrak S, Bellanova G, Beltran MA, Bini R, Boal M, Borodach AV, Bouliaris K, Branger F, Brunelli D, Catani M, Che Jusoh A, Chichom-Mefire A, Cocorullo G, Colak E, Costa D, Costa S, Cui Y, Curca GL, Curry T, Das K, Delibegovic S, Demetrashvili Z, Di Carlo I, Drozdova N, El Zalabany T, Enani MA, Faro M, Gachabayov M, Gimenez Maurel T, Gkiokas G, Gomes CA, Gonsaga RA, Guercioni G, Guner A, Gupta S, Gutierrez S, Hutan M, Ioannidis O, Isik A, Izawa Y, Jain SA, Jokubauskas M, Karamarkovic A, Kauhanen S, Kaushik R, Kenig J, Khokha V, Kim JI, Kong V, Koshy R, Krasniqi A, Kshirsagar A, Kuliesius Z, Lasithiotakis K, Leao P, Lee JG, Leon M, Lizarazu Perez A, Lohsiriwat V, Lopez-Tomassetti Fernandez E, Lostoridis E, Mn R, Major P, Marinis A, Marrelli D, Martinez-Perez A, Marwah S, McFarlane M, Melo RB, Mesina C, Michalopoulos N, Moldovanu R, Mouaqit O, Munyika A, Negoi I, Nikolopoulos I, Nita GE, Olaoye I, Omari A, Ossa PR, Ozkan Z, Padmakumar R, Pata F, Pereira Junior GA, Pereira J, Pintar T, Pouggouras K, Prabhu V, Rausei S, Rems M, Rios-Cruz D, Sakakushev B, Sanchez de Molina ML, Seretis C, Shelat V, Simoes RL, Sinibaldi G, Skrovina M, Smirnov D, Spyropoulos C, Tepp J, Tezcaner T, Tolonen M, Torba M, Ulrych J, Uzunoglu MY, van Dellen D, van Ramshorst GH, Vasquez G, Venara A, Vereczkei A, Vettoretto N, Vlad N, Yadav SK, Yilmaz TU, Yuan KC, Zachariah SK, Zida M, Zilinskas J, Ansaloni L. Global validation of the WSES Sepsis Severity Score for patients with complicated intra-abdominal infections: a prospective multicentre study (WISS Study). World J Emerg Surg. 2015 Dec 16;10:61. doi: 10.1186/s13017-015-0055-0. eCollection 2015. PMID 26677396
- [Result] Sartelli M, Abu-Zidan FM, Ansaloni L, Bala M, Beltran MA, Biffl WL, Catena F, Chiara O, Coccolini F, Coimbra R, Demetrashvili Z, Demetriades D, Diaz JJ, Di Saverio S, Fraga GP, Ghnnam W, Griffiths EA, Gupta S, Hecker A, Karamarkovic A, Kong VY, Kafka-Ritsch R, Kluger Y, Latifi R, Leppaniemi A, Lee JG, McFarlane M, Marwah S, Moore FA, Ordonez CA, Pereira GA, Plaudis H, Shelat VG, Ulrych J, Zachariah SK, Zielinski MD, Garcia MP, Moore EE. The role of the open abdomen procedure in managing severe abdominal sepsis: WSES position paper. World J Emerg Surg. 2015 Aug 12;10:35. doi: 10.1186/s13017-015-0032-7. eCollection 2015. PMID 26269709
- [Result] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Result] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Intensive Care Med. 2008 Jan;34(1):17-60. doi: 10.1007/s00134-007-0934-2. Epub 2007 Dec 4. PMID 18058085
- [Result] Slade E, Tamber PS, Vincent JL. The Surviving Sepsis Campaign: raising awareness to reduce mortality. Crit Care. 2003 Feb;7(1):1-2. doi: 10.1186/cc1876. Epub 2003 Jan 8. PMID 12617727
- [Result] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Derived] Kirkpatrick AW, Coccolini F, Tolonen M, Minor S, Catena F, Gois E Jr, Doig CJ, Hill MD, Ansaloni L, Chiarugi M, Tartaglia D, Ioannidis O, Sugrue M, Colak E, Hameed SM, Lampela H, Agnoletti V, McKee JL, Garraway N, Sartelli M, Ball CG, Parry NG, Voght K, Julien L, Kroeker J, Roberts DJ, Faris P, Tiruta C, Moore EE, Ammons LA, Anestiadou E, Bendinelli C, Bouliaris K, Carroll R, Ceresoli M, Favi F, Gurrado A, Rezende-Neto J, Isik A, Cremonini C, Strambi S, Koukoulis G, Testini M, Trpcic S, Pasculli A, Picariello E, Abu-Zidan F, Adeyeye A, Augustin G, Alconchel F, Altinel Y, Hernandez Amin LA, Aranda-Narvaez JM, Baraket O, Biffl WL, Baiocchi GL, Bonavina L, Brisinda G, Cardinali L, Celotti A, Chaouch M, Chiarello M, Costa G, de'Angelis N, De Manzini N, Delibegovic S, Di Saverio S, De Simone B, Dubuisson V, Fransvea P, Garulli G, Giordano A, Gomes C, Hayati F, Huang J, Ibrahim AF, Huei TJ, Jailani RF, Khan M, Luna AP, Malbrain MLNG, Marwah S, McBeth P, Mihailescu A, Morello A, Mulita F, Murzi V, Mohammad AT, Parmar S, Pak A, Wong MP, Pantalone D, Podda M, Puccioni C, Rasa K, Ren J, Roscio F, Gonzalez-Sanchez A, Sganga G, Scheiterle M, Slavchev M, Smirnov D, Tosi L, Trivedi A, Vega JAG, Waledziak M, Xenaki S, Winter D, Wu X, Zakaria AD, Zakaria Z. The unrestricted global effort to complete the COOL trial. World J Emerg Surg. 2023 May 11;18(1):33. doi: 10.1186/s13017-023-00500-z. PMID 37170123
- [Derived] Ng-Kamstra JS, Rennert-May E, McKee J, Lundgren S, Manns B, Kirkpatrick AW. Protocol for a parallel economic evaluation of a trial comparing two surgical strategies in severe complicated intra-abdominal sepsis: the COOL-cost study. World J Emerg Surg. 2020 Feb 21;15(1):15. doi: 10.1186/s13017-020-00294-4. PMID 32085778
- [Derived] Doig CJ, Page SA, McKee JL, Moore EE, Abu-Zidan FM, Carroll R, Marshall JC, Faris PD, Tolonen M, Catena F, Cocolini F, Sartelli M, Ansaloni L, Minor SF, Peirera BM, Diaz JJ, Kirkpatrick AW; Closed Or Open after Laparotomy (COOL) after Source Control for Severe Complicated Intra-Abdominal Sepsis Investigators. Ethical considerations in conducting surgical research in severe complicated intra-abdominal sepsis. World J Emerg Surg. 2019 Aug 5;14:39. doi: 10.1186/s13017-019-0259-9. eCollection 2019. PMID 31404221
- [Derived] Kirkpatrick AW, Coccolini F, Ansaloni L, Roberts DJ, Tolonen M, McKee JL, Leppaniemi A, Faris P, Doig CJ, Catena F, Fabian T, Jenne CN, Chiara O, Kubes P, Manns B, Kluger Y, Fraga GP, Pereira BM, Diaz JJ, Sugrue M, Moore EE, Ren J, Ball CG, Coimbra R, Balogh ZJ, Abu-Zidan FM, Dixon E, Biffl W, MacLean A, Ball I, Drover J, McBeth PB, Posadas-Calleja JG, Parry NG, Di Saverio S, Ordonez CA, Xiao J, Sartelli M; Closed Or Open after Laparotomy (COOL) after Source Control for Severe Complicated Intra-Abdominal Sepsis Investigators. Closed Or Open after Source Control Laparotomy for Severe Complicated Intra-Abdominal Sepsis (the COOL trial): study protocol for a randomized controlled trial. World J Emerg Surg. 2018 Jun 22;13:26. doi: 10.1186/s13017-018-0183-4. eCollection 2018. PMID 29977328
- [Derived] Tolonen M, Coccolini F, Ansaloni L, Sartelli M, Roberts DJ, McKee JL, Leppaniemi A, Doig CJ, Catena F, Fabian T, Jenne CN, Chiara O, Kubes P, Kluger Y, Fraga GP, Pereira BM, Diaz JJ, Sugrue M, Moore EE, Ren J, Ball CG, Coimbra R, Dixon E, Biffl W, MacLean A, McBeth PB, Posadas-Calleja JG, Di Saverio S, Xiao J, Kirkpatrick AW; From the Closed Or Open after Laparotomy (COOL) for Source Control in Severe Complicated Intra-Abdominal Sepsis Investigators. Getting the invite list right: a discussion of sepsis severity scoring systems in severe complicated intra-abdominal sepsis and randomized trial inclusion criteria. World J Emerg Surg. 2018 Apr 6;13:17. doi: 10.1186/s13017-018-0177-2. eCollection 2018. PMID 29636790